CLINICAL TRIAL: NCT01680133
Title: Regulation of Lipolysis by Insulin in Skeletal Muscle and Adipose Tissue in Type 2 Diabetes
Brief Title: Regulation of Tissue Lipolysis by Insulin in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Other Study IDs: 07-3-037; 91611074 (Other Grant/Funding Number: The Netherlands Organisation for Scientific Research)
Record Dates: First submitted 2012-08-21; First posted 2012-09-07 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — adipose tissue and skeletal muscle biopsies

GROUPS / COHORTS (2):
- NGT: Normal glycaemic healthy control men, age between 45-65, BMI 25-35 kg/m2
  Interventions: Other: Hyperinsulinemic euglycemic clamp
- T2D: Type 2 diabetic men, age 45-65 yrs, BMI 25-35, diagnosed >5yrs and Hba1c 7-9%
  Interventions: Other: Hyperinsulinemic euglycemic clamp

INTERVENTIONS:
Other: Hyperinsulinemic euglycemic clamp

SUMMARY:
Inadequate suppression of intramuscular and adipose tissue lipolysis, and consequent excessive delivery of fatty acids to ectopic tissues (e.g. muscle, pancreas and liver) could play an important role in the development and exacerbating of insulin resistance. Therefore, the investigators propose to study the regulation of adipose tissue and skeletal muscle lipolysis, as well as further characterize the intracellular lipolytic pathways within these tissues, in obese normoglycaemic versus long-term diagnosed type 2 diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Normal blood pressure (SBP 100-140 mmHg, DBP 60-90 mmHg)
* weight stable in last 3 months

Exclusion Criteria:

* Smokers
* people with intensive fitness training (e.g. athletes > 3 times/week)
* History of cardiovascular diseases
* Bleeding disorders
* Use of medication interfering with the study endpoints/hypotheses (e.g. beta-blockers)
* Not to be able to understand the study information
* Subjects on a special diet or vegetarian
* Blood donation 2 months prior to the study and during the study
* Participating in an other study

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normoglycemic men and type 2 diabetic men
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity of adipose tissue and skeletal muscle lipolysis | 8, 20 and 40 mU insulin (2 hours)
  Changes from baseline in glycerol (lactate, pyruvate and glucose) in tissue microdialysate during a 3 step euglycemic hyperinsulinemic clamp (8, 20 and 40mU of insulin), every step for 2h

SECONDARY OUTCOMES:
Baseline adipose tissue and skeletal muscle gene expression | baseline
  gene expression of genes related to lipid, glucose metabolism, insulin signalling will be measured in baseline adipose tissue and skeletal muscle biopsies
Baseline skeletal muscle lipid accumulation | Baseline
  Baseline skeletal muscle lipid accumulation is measured (TAG, DAG, Phospholipid and fatty acids)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Blaak, PhD, Principal Investigator — Maastricht University Medical centre
Locations (1):
- Department of Human Biology, Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Background] Jocken JW, Moro C, Goossens GH, Hansen D, Mairal A, Hesselink MK, Langin D, van Loon LJ, Blaak EE. Skeletal muscle lipase content and activity in obesity and type 2 diabetes. J Clin Endocrinol Metab. 2010 Dec;95(12):5449-53. doi: 10.1210/jc.2010-0776. Epub 2010 Sep 15. PMID 20843949
- [Background] Jocken JW, Roepstorff C, Goossens GH, van der Baan P, van Baak M, Saris WH, Kiens B, Blaak EE. Hormone-sensitive lipase serine phosphorylation and glycerol exchange across skeletal muscle in lean and obese subjects: effect of beta-adrenergic stimulation. Diabetes. 2008 Jul;57(7):1834-41. doi: 10.2337/db07-0857. Epub 2008 Apr 8. PMID 18398140
- [Background] Jocken JW, Goossens GH, van Hees AM, Frayn KN, van Baak M, Stegen J, Pakbiers MT, Saris WH, Blaak EE. Effect of beta-adrenergic stimulation on whole-body and abdominal subcutaneous adipose tissue lipolysis in lean and obese men. Diabetologia. 2008 Feb;51(2):320-7. doi: 10.1007/s00125-007-0866-y. Epub 2007 Dec 5. PMID 18060661
- [Background] Boon H, Blaak EE, Saris WH, Keizer HA, Wagenmakers AJ, van Loon LJ. Substrate source utilisation in long-term diagnosed type 2 diabetes patients at rest, and during exercise and subsequent recovery. Diabetologia. 2007 Jan;50(1):103-12. doi: 10.1007/s00125-006-0482-2. Epub 2006 Nov 28. PMID 17131144
- [Derived] Jocken JW, Goossens GH, Boon H, Mason RR, Essers Y, Havekes B, Watt MJ, van Loon LJ, Blaak EE. Insulin-mediated suppression of lipolysis in adipose tissue and skeletal muscle of obese type 2 diabetic men and men with normal glucose tolerance. Diabetologia. 2013 Oct;56(10):2255-65. doi: 10.1007/s00125-013-2995-9. Epub 2013 Aug 2. PMID 23907381